CLINICAL TRIAL: NCT01318525
Title: A Multicentre, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and the Safety of ALF-5755 in Patients With Nonacetaminophen Severe Acute Hepatitis and Early Stage Acute Liver Failure
Brief Title: Efficacy & Safety of ALF-5755 in Patients With Nonacetaminophen Severe Acute Hepatitis & Early Stage Acute Liver Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alfact Innovation (Industry)
Responsible Party: Paul Amouyal, Alfact Innovation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALF-5755_P2_ALF
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Liver Failure, Acute
MeSH Terms: conditions — Liver Failure, Acute | interventions — ALF-5755; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALF-5755 (Experimental)
  Interventions: Drug: ALF-5755
- Saline solution (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Saline solution (0.9% NaCl)

INTERVENTIONS:
Drug: ALF-5755 — 10 mg (25 ml) given in slow intravenous infusion over 10 minutes with an automatic syringe
  Arms: ALF-5755
Drug: Saline solution (0.9% NaCl) — 25 ml given in slow intravenous infusion over 10 minutes with an automatic syringe
  Arms: Saline solution (0.9% NaCl)

SUMMARY:
Acute liver failure is a rare but dramatic disease, often affecting young people, marked by the sudden loss of liver function in a person without preexisting liver disease.

ALF-5755 has been shown to promote cell survival after apoptotic or oxidative stress, and liver cell regeneration in primary cultures and in vivo. ALF-5755 may become, in this dramatic disease with high unmet medical need, a future therapy for the treatment of patients suffering from severe acute hepatitis (SAH) and acute liver failure (ALF) not due to acetaminophen overdose, where liver transplantation is the sole treatment in the absence of spontaneous recovery.

The primary objective of the study is to evaluate the efficacy of ALF-5755 versus placebo.

A minimum of 60 patients will be recruited into the study in the following two treatment groups:

* Group A: approximately 30 patients will receive ALF-5755
* Group B: approximately 30 patients will receive placebo (physiological saline solution: 0.9% NaCl)

Patients will receive 10 mg (25 ml) of ALF5755 or placebo every 12 hours over 3 days in slow intravenous infusions over 10 minutes using automatic syringes.

ELIGIBILITY:
Inclusion Criteria:

* A signed written informed consent from patient or from patient's next of kin or from an authorized person according to local procedures
* Early stage acute liver failure OR severe acute hepatitis defined as:
* 15% ≤ PR < 50%
* No hepatic encephalopathy, OR grade I or II encephalopathy (Appendix E)
* Presumed acute illness onset of less than 26 weeks
* No evidence of underlying chronic liver disease
* Patient who can receive first treatment dose within the first 48 hours after biological baseline assessment
* Age ≥ 18 and ≤ 65 years
* Contraception (only for females of childbearing potential) to be taken throughout the study until D21. Sole mechanic contraceptives, such as condoms, are advised. Note: Oral contraceptives may have contraindications in case of severe acute hepatitis and acute liver failure
* Patient affiliated to social security insurance system.

Exclusion Criteria:

* Acetaminophen-induced hepatitis defined as acetaminophen intake > 4 g/day, at least once in the 7 days prior to baseline
* Shock liver (ischemic hepatopathy) OR HELLP syndrome OR Budd-Chiari syndrome OR intrahepatic malignancy
* Serum creatinine ≥ 180 μmol/L
* Body Mass Index (BMI) ≥ 35
* Septic shock requiring administration of inotropic drugs
* Uncontrolled active bleeding
* Patients who received fresh frozen plasma, PPSB (Prothrombin-Proconvertin-Stuart-B), or vitamin K infusion over the last 48 hours
* Patient receiving liver support device treatment, including but not exclusively bioartificial liver (BAL), Extracorporeal Liver Assist Device (ELAD), transgenic pig perfusion
* Patient receiving hemodialysis, hemofiltration or hemodiafiltration treatment
* Intractable arterial hypotension (arterial systolic blood pressure equal to or below 70 mmHg) present or require inotropic drugs at baseline
* Human Immunodeficiency Virus (HIV) positive patient
* Active cancer
* Pregnancy or breast-feeding
* Surgery within 4 weeks prior to baseline, or unsolved surgical disease outside liver transplantation.
* Patient included in another clinical trial within 4 weeks prior to baseline
* Patient with organ or bone-marrow allograft
* Absolute contra-indication to liver transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-05 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Rate of change of Prothrombin Rate initiation | Over a period of 72 hours from baseline

SECONDARY OUTCOMES:
Rate of change of Factor V (FV) plasma level | Over a period of 72 hours from baseline
Rate of change of international normalized ratio (INR) | Over a period of 72 hours from baseline
Rate of change of alanine transaminases (ALT) plasma level | Over a period of 72 hours from baseline
Rate of change of aspartate transaminases (AST) plasma level | Over a period of 72 hours from baseline
Change of Hepatic Encephalopathy Grade (HE grade) | Over a period of 72 hours from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul Amouyal, Study Director — Alfact Innovation
Locations (12):
- France (12):
  - CHU de Besançon, Besançon
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHU de Grenoble, Grenoble
  - Hôpital Claude Huriez, Lille
  - Hôpital Croix-Rousse, Lyon
  - Hôpital Conception, Marseille
  - Hôpital Saint-Eloi, Montpellier
  - Hôpital de l'Archet 2, Nice
  - Hôpital Saint Antoine, Paris
  - Hôpital La Pitié Salpétrière, Paris
  - Centre Hépatobiliaire Paul Brousse, Villejuif

REFERENCES:
- [Background] Christa L, Felin M, Morali O, Simon MT, Lasserre C, Brechot C, Seve AP. The human HIP gene, overexpressed in primary liver cancer encodes for a C-type carbohydrate binding protein with lactose binding activity. FEBS Lett. 1994 Jan 3;337(1):114-8. doi: 10.1016/0014-5793(94)80640-3. PMID 8276102
- [Background] Hoofnagle JH, Carithers RL Jr, Shapiro C, Ascher N. Fulminant hepatic failure: summary of a workshop. Hepatology. 1995 Jan;21(1):240-52. PMID 7806160
- [Background] Iovanna JL, Dagorn JC. The multifunctional family of secreted proteins containing a C-type lectin-like domain linked to a short N-terminal peptide. Biochim Biophys Acta. 2005 May 25;1723(1-3):8-18. doi: 10.1016/j.bbagen.2005.01.002. Epub 2005 Jan 21. PMID 15715980
- [Background] Kondo T, Suda T, Fukuyama H, Adachi M, Nagata S. Essential roles of the Fas ligand in the development of hepatitis. Nat Med. 1997 Apr;3(4):409-13. doi: 10.1038/nm0497-409. PMID 9095174
- [Background] Lasserre C, Christa L, Simon MT, Vernier P, Brechot C. A novel gene (HIP) activated in human primary liver cancer. Cancer Res. 1992 Sep 15;52(18):5089-95. PMID 1325291
- [Background] Lieu HT, Batteux F, Simon MT, Cortes A, Nicco C, Zavala F, Pauloin A, Tralhao JG, Soubrane O, Weill B, Brechot C, Christa L. HIP/PAP accelerates liver regeneration and protects against acetaminophen injury in mice. Hepatology. 2005 Sep;42(3):618-26. doi: 10.1002/hep.20845. PMID 16116631
- [Background] Lieu HT, Simon MT, Nguyen-Khoa T, Kebede M, Cortes A, Tebar L, Smith AJ, Bayne R, Hunt SP, Brechot C, Christa L. Reg2 inactivation increases sensitivity to Fas hepatotoxicity and delays liver regeneration post-hepatectomy in mice. Hepatology. 2006 Dec;44(6):1452-64. doi: 10.1002/hep.21434. PMID 17133485
- [Background] Polson J, Lee WM; American Association for the Study of Liver Disease. AASLD position paper: the management of acute liver failure. Hepatology. 2005 May;41(5):1179-97. doi: 10.1002/hep.20703. No abstract available. PMID 15841455
- [Background] Simon MT, Pauloin A, Normand G, Lieu HT, Mouly H, Pivert G, Carnot F, Tralhao JG, Brechot C, Christa L. HIP/PAP stimulates liver regeneration after partial hepatectomy and combines mitogenic and anti-apoptotic functions through the PKA signaling pathway. FASEB J. 2003 Aug;17(11):1441-50. doi: 10.1096/fj.02-1013com. PMID 12890698
- [Derived] Nalpas B, Ichai P, Jamot L, Carbonell N, Rudler M, Mathurin P, Durand F, Gerken G, Manns M, Trautwein C, Larrey D, Radenne S, Duvoux C, Leroy V, Bernuau J, Faivre J, Moniaux N, Brechot C, Amouyal G, Amouyal P, Samuel D. A Proof of Concept, Phase II Randomized European Trial, on the Efficacy of ALF-5755, a Novel Extracellular Matrix-Targeted Antioxidant in Patients with Acute Liver Diseases. PLoS One. 2016 Mar 16;11(3):e0150733. doi: 10.1371/journal.pone.0150733. eCollection 2016. PMID 26983031